CLINICAL TRIAL: NCT00716833
Title: Etoricoxibe - Preemptive and Postoperative Analgesia for Abdominal and Thoracic Surgery
Acronym: EPPA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dominik Irnich, PD Dr. Dominik Irnich, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MPC-UM-0002-DI
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Pain; Abdominal Surgery; Thoracic Surgery
Keywords: pain; coxibe; preemptive; abdominothoracic; sensibilisation; Analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preemptive (Active Comparator): Preemptive group patients get Etoricoxibe twice (before and after surgery) or just a single preoperative dose
  Interventions: Drug: Etoricoxibe
- Postoperative (Placebo Comparator): Postoperative group patients get placebo before surgery and either a drug application or a placebo again after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etoricoxibe — Preemptive group patients get Etoricoxibe either twice (before and after surgery) or just a single preoperative dose.
  Other Names: Etoricoxibe 120mg Registration-N° 59863.02.00
  Arms: Preemptive
Drug: Placebo — Postoperative group patients get placebo before surgery and either a drug application or a placebo again after surgery (so called 2x2 factorial study design).
  Other Names: Placebo-Etoricoxibe
  Arms: Postoperative

SUMMARY:
This randomised placebo controlled double-blinded bicentre study (phase III) was designed to evaluate the preemptive and postoperative analgetic impact of etoricoxibe in open abdominal and thoracic surgery. Etoricoxib selectively inhibits isoform 2 of cyclo-oxigenase enzyme (COX-2).

Therefore 120 patients (ASA-risk 1-2) with upcoming abdominal or thoracic surgery should be included into this study. Patients are randomly allocated to either the preemptive or the postoperative Etoricoxibe group. These two groups are divided each into two arms. Preemptive group patients get Etoricoxibe either twice (before and after surgery) or just a single preoperative dose. Postoperative group patients get placebo before surgery and either a drug application or a placebo again after surgery (so called 2x2 factorial study design).

Cumulative use of morphine as assessed within first 48 hours after surgery is the primary trial outcome indicating the analgesic potency of Etoricoxibe.

In addition, changes in patients level of sensibilisation will be measured with help of quantitative sensory testing (a standardised procedure) before and after surgery (secondary outcome). In addition pharmacogenetic testing will provide information about genetic aberrations (so called polymorphisms) of the patients enzymes that should be compared to the individual reaction regarding Etoricoxibe.

The results will give hint about the analgesic impact of etoricoxibe in acute postoperative pain. There will be findings for preemptive analgesia and nerval processes. All this could lead to an improvement of postoperative pain relief while administrating preemptively a COX-2 selective inhibitor before surgery.

DETAILED DESCRIPTION:
Etoricoxib (brand name Arcoxia worldwide; also Algix and Tauxib in Italy) is a new COX-2 selective inhibitor (approx. 106.0 times more selective for COX-2 inhibition over COX-1). Doses are 120 mg/day for acute pain. Current therapeutic indications are: treatment of rheumatoid arthritis, osteoarthritis, ankylosing spondylitis, chronic low back pain, acute pain and gout. Note that approved indications differ by country.

Like any other COX-2 selective inhibitor, Etoricoxib selectively inhibits isoform 2 of cyclo-oxigenase enzyme (COX-2). This reduces the generation of prostaglandins (PGs) from arachidonic acid. Among the different functions exerted by PGs, their role in the inflammation cascade should be highlighted. COX-2 selective inhibitor (aka "COXIB") showed less marked activity on type 1 cycloxigenase compared to traditional non-steroidal anti-inflammatory drugs (NSAID). This reduced activity is the cause of reduced gastrointestinal toxicity.

Quantitative sensory tests (QST) are techniques employed to measure the intensity of stimuli needed to produce specific sensory perceptions. They are used to evaluate a sensory detection threshold or other sensory responses from supra-threshold stimulation. The common physical stimuli are (i) touch-pressure, (ii) vibration, and (iii) coolness, warmth, cold pain, and heat pain. In QST, the subject must be able to comprehend what is being asked by the test, alert and not taking mind-altering medications, and not biased to a certain test outcome.

ELIGIBILITY:
Inclusion Criteria:

* Programmed abdominal or thoracic surgery
* Patients > 18 yrs
* Patients are aware of German language
* Participation is voluntary
* ASA-risk class 1-2 (American Society of Anesthesiologists guidelines)

Exclusion Criteria:

* Severe cardiac, pulmonary, renal or neurologic disease
* ASA risk III and IV
* Insulin dependent Diabetes mellitus
* Polyneuropathy
* Chronic pain
* Use of analgesic drugs
* Ulcus duodeni
* Ulcus ventriculi
* Time after intestinal bleeding
* Allergy reactions towards coxibes or coxibe-like drugs
* Pregnancy and lactation
* Severe hepatic disease (Albumin < 25 g/l or Child-Pugh-Score ≥ 10)
* Children and Teenager < 16 years
* Chronic intestinal inflammation
* Heart failure (NYHA II - IV)
* Inbalancend arterial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-02; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cumulative use of morphine as assessed within first 48 hours after surgery | first 48 hours

SECONDARY OUTCOMES:
Changes in patients level of sensibilisation will be measured with help of quantitative sensory testing (a standardised procedure) before and after surgery. | preoperative and 48h postoperative
Pharmacogenetic testing will provide information about genetic aberrations (so called polymorphisms) of the patients enzymes that should be compared to the individual reaction regarding Etoricoxibe. | 48 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Irnich, PD. Dr., Principal Investigator — Multidisciplinary Pain Centre, Department of Anaesthesiology, University of Munich, Munich, Germany
Locations (2):
- Germany (2):
  - Zentrum für Pneumologie und Thoraxchirurgie, Asklepios Fachkliniken München-Gauting, Gauting
  - Chirurgische Klinik und Poliklinik, Innenstadt, Klinikum der Universität München, München

REFERENCES:
- [Background] Fleckenstein J, Kramer S, Offenbacher M, Schober G, Plischke H, Siebeck M, Mussack T, Hatz R, Lehmeyer L, Lang PM, Heindl B, Conzen P, Irnich D. Etoricoxib--preemptive and postoperative analgesia (EPPA) in patients with laparotomy or thoracotomy--design and protocols. Trials. 2010 May 27;11:66. doi: 10.1186/1745-6215-11-66. PMID 20504378
- [Derived] Fleckenstein J, Kohls N, Evtouchenko E, Lehmeyer L, Kramer S, Lang PM, Siebeck M, Mussack T, Hatz R, Heindl B, Conzen P, Rehm M, Czerner S, Zwissler B, Irnich D. No effect of the cyclooxygenase-2 inhibitor etoricoxib on pre-emptive and post-operative analgesia in visceral surgery: results of a randomized controlled trial. Eur J Pain. 2016 Feb;20(2):186-95. doi: 10.1002/ejp.699. Epub 2015 Mar 31. PMID 25828692